CLINICAL TRIAL: NCT00131170
Title: Paravertebral Block for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PVB1
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: paravertebral block

SUMMARY:
The effect of paravertebral block in combination with general anaesthesia is studied in a double blind fashion.

DETAILED DESCRIPTION:
Patients having surgery for breast cancer receive a paravertebral blockade at C8-Th4 with either Naropin 0.5% or saline. General anaesthesia is then provided with laryngeal mask intubation, propofol infusion and fentanyl i.v. as needed. The effect on postoperative pain ([VAS] and fentanyl PCA doses taken) and postoperative nausea and vomiting is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Breast surgery

Exclusion Criteria:

* Infections
* Coagulation disorder
* Allergy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Nausea and vomiting 2 hours postoperatively, and 1 and 2 days postoperatively | 2 days

SECONDARY OUTCOMES:
Dosage of analgesic | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Palle Carlsson, MD Dr Sci, Principal Investigator — Dept anesthesiology, Arhus University Hospital
Locations (1):
- Dept of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark